CLINICAL TRIAL: NCT07057089
Title: Clinical Exploration of Involved-field Radiotherapy-TNT Combined With PD-1 Inhibitor for pMMR Locally Advanced Rectal Cancer: a Prospective, Open-label, Randomized Controlled Trial (Neo-Field I)
Brief Title: Involved-field Radiotherapy-TNT Combined With PD-1 Inhibitor for pMMR Locally Advanced Rectal Cancer (Neo-Field I)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARK-Rectal cancer-001
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Capecitabine; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Involve-field radiotherapy-TNT+Camrelizumab (Experimental): Patients received Involve-field radiotherapy (25Gy/5f, including the primary rectal tumor, metastatic or suspected pelvic lymph nodes, mesorectal, and presacral regions). Four cycles of CAPOX plus Carilizumab were given to patients 1-2 weeks after chemoradiotherapy completion.
  Patients were evaluated 2-3 weeks after the end of treatment. Patients who met the cCR criteria could choose to undergo surgical treatment or not. For patients who did not meet the cCR criteria, surgical treatment was recommended. For patients who refused surgery, the patients in the trial group continued to receive 4 cycles of CAPOX chemotherapy combined with camrelizumab.
  Interventions: Drug: Camrelizumab; Drug: CAPOX; Radiation: Involve-field irradiation; Procedure: TME surgery
- Elective nodal irradiation-TNT (Other): Patients received elective nodal long-course concurrent chemoradiotherapy (50.4 Gy/28f). Capecitabine (825 mg/m² bid) was administered orally on radiotherapy days. Four cycles of CAPOX were given to patients 1-2 weeks after chemoradiotherapy completion.
  Patients were evaluated 2-3 weeks after the end of treatment. Patients who met the cCR criteria could choose to undergo surgical treatment or not. For patients who did not meet the cCR criteria, surgical treatment was recommended. For patients who refused surgery, the patients in the trial group continued to receive 4 cycles of CAPOX chemotherapy.
  Interventions: Drug: Capecitabine; Drug: CAPOX; Radiation: Elective nodal irradiation; Procedure: TME surgery

INTERVENTIONS:
Drug: Capecitabine — Capecitabine: 825mg/m2, bid;
  Arms: Elective nodal irradiation-TNT
Drug: Camrelizumab — Camrelizumab: 200mg
  Arms: Involve-field radiotherapy-TNT+Camrelizumab
Drug: CAPOX — CAPOX
Radiation: Involve-field irradiation — Involve-field irradiation: Primary rectal tumor + metastatic or suspicious pelvic lymph nodes, mesorectal region, and presacral region
  Arms: Involve-field radiotherapy-TNT+Camrelizumab
Radiation: Elective nodal irradiation — Elective nodal irradiation: Large pelvic field
  Arms: Elective nodal irradiation-TNT
Procedure: TME surgery — TME surgery

SUMMARY:
The purpose of this study is to explore the efficacy and safety of involved-field radiotherapy-TNT combined with PD-1 inhibitors in pMMR locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. Pathologic diagnosis of adenocarcinoma of the rectum, definite pMMR type;
4. Clinical staging of T3-4NanyM0 or T1-2N+M0 (based on AJCC 8th edition staging criteria);
5. The lower margin of the primary tumor is located below the peritoneal reflex or the lower margin of the tumor is ≤10 cm from the anal verge;
6. Pre-enrollment laboratory indicators meet the following indicator ranges： 1)Blood: absolute neutrophils ≥1.5×10^9/L, platelets ≥100×10^9/L, hemoglobin ≥90g/L; 2)Liver and kidney function: ALT/AST ≤ 2.5 x ULN, total bilirubin ≤ 1.5 x ULN, creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 60mL/min (Cockcroft-Gault formula)； 3)Coagulation: INR ≤ 1.5, APTT ≤ 1.5 x ULN (for those not receiving anticoagulation)；
7. Women or men of childbearing potential need to agree to use effective contraception during the study and for 6 months after the last treatment session;
8. Voluntary written informed consent and commitment to complete the full treatment and follow-up program.

Exclusion Criteria:

1. Pathologic type is other specific types such as neuroendocrine carcinoma, squamous carcinoma, etc;
2. Previous radiotherapy, chemotherapy, targeted or immunotherapy for rectal cancer;
3. Active autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis requiring long-term immunosuppressive therapy)；
4. Presence of active infection (e.g. HIV, HBV/HCV viral load positive requiring stabilization on antiretroviral therapy)；
5. Severe cardiovascular disease (e.g., myocardial infarction within 6 months, unstable angina, uncontrolled hypertension >160/100 mmHg)；
6. History of other malignant tumors (except non-melanoma skin cancers, cervical cancer in situ, etc. cured for ≥5 years)；
7. Uncontrolled diabetes mellitus (HbA1c > 8%), abnormal thyroid function (TSH outside normal range and requiring pharmacologic intervention)；
8. Severe chronic bowel disease (e.g., Crohn's disease, active ulcerative colitis)； Patients deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
CR rate | within 5 weeks
  CR defined as patient achieving pCR and cCR.

SECONDARY OUTCOMES:
MPR rate | within 3 weeks after surgery
  MPR defined as patients achieving a major pathological response after surgery.
R0-resection rate | within 3 weeks after surgery
  R0-resection defined as patients without tumor cell infiltration in the tissue 1mm from the resection margin
Preservation rate of adjacent invaded organs | within 3 weeks after surgery
  The involved organs were successfully preserved during the operation
ORR | within 5 weeks
  Defined as the percentage of complete response (CR) and partial response (PR) to tumor volume reduction according to RECIST v1.1 criteria
3-year Event Free Survival | 3 years
  EFS defined as time from randomization to objectively observed tumor progression (local recurrence, new disease, or distant metastasis), development of a second malignancy, or death (death from any cause).
3-year OS | 3 years
  OS defined as time from randomization to death from any cause.
Incidence of adverse reactions | 1 year
  Occurrence of adverse reactions during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Fengpeng Wu, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, China

IPD SHARING:
Plan to Share IPD: Undecided